CLINICAL TRIAL: NCT07333872
Title: Evaluation of Pulpotomy, Partial Pulpotomy, and Direct Pulp Capping Using Mineral Trioxide Aggregate in Primary Molars. A Randomized Clinical Trial.
Brief Title: Evaluation of Pulpotomy, Partial Pulpotomy, and Direct Pulp Capping Using Mineral Trioxide Aggregate.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DU:025052113
Record Dates: First submitted 2026-01-01; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: Vital Pulp Therapy in Primary Teeth
MeSH Terms: interventions — Dental Pulp Capping; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct pulp capping (Experimental): Technique of vital pulp therapy to cap pin point exposure
  Interventions: Procedure: pulp capping with MTA
- Partial pulpotomy (Experimental): Technique of vital pulp therapy to cap widened pulp exposure
  Interventions: Procedure: pulp capping with MTA
- Pulpotomy (Experimental): Technique of vital pulp therapy of capping radicular pulp after removal of coronal pulp
  Interventions: Procedure: pulp capping with MTA

INTERVENTIONS:
Procedure: pulp capping with MTA — Capping of the pulp tissue with a biocompatible material (MTA)

SUMMARY:
A comparative evaluation for three vital pulp therapy techniques in primary molars using the same material (MTA)

ELIGIBILITY:
Inclusion Criteria:

* articipants were cooperative children (4-7 years) with no systemic diseases or relevant allergies. Eligible teeth were restorable primary second molars with deep carious lesions and a diagnosis of reversible pulpitis,

Exclusion Criteria:

* spontaneous pain, edema, fistula, pathological mobility, or percussion sensitivity.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Spontaneous pain | 12 months
  numeric rating scale (presence or abscence of pain) 0 is best result 10 is the worst
Radiolucency of the periapical or furcation area | Follow up for 12 months
  measuring tool is x-ray

SECONDARY OUTCOMES:
Presence or absence of fistula | 12 months
  Visual inspection
Pathological mobility | 12 months
  Graded clinical by applying pressure by end of mirror
Sensitivity on percussion | 12 months
  Methods of tapping on surface in clinical examination
Widening of personal ligament space | 12 months
  Measuring tool is xray
Internal or e ternal resorption | 12 months
  Measuring tool is xray

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university for science and technology, Gamasa, Dakahlia Governorate, Egypt